CLINICAL TRIAL: NCT05995704
Title: A Phase 1, Randomized, Placebo-Controlled, Double-Blind, Single Center, Multiple-Dose, Parallel Trial Evaluating the Impact of Apraglutide on Gastric Emptying of Liquids in Healthy Subjects
Brief Title: Evaluation of Apraglutide on Gastric Emptying
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: VectivBio AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: TA799-020
Record Dates: First submitted 2023-02-22; First posted 2023-08-16 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-01

CONDITIONS: Healthy Subjects
Keywords: Gastric emptying; Pharmacokinetics of acetaminophen
MeSH Terms: interventions — apraglutide; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The pharmacist and designated staff will be unblinded.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Apraglutide SC injections (Experimental)
  Interventions: Drug: Apraglutide; Drug: Acetaminophen
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: Acetaminophen

INTERVENTIONS:
Drug: Apraglutide — Peptide analogue of GLP-2
  Arms: Apraglutide SC injections
Drug: Placebo — Matching placebo to apraglutide
  Arms: Placebo
Drug: Acetaminophen — Acetaminophen mixed with a liquid meal

SUMMARY:
The primary objective is to assess the effect of apraglutide on gastric emptying of liquids in healthy subjects, as measured by the PK of acetaminophen mixed with a liquid meal.

DETAILED DESCRIPTION:
This is a single-center, double-blind, randomized, multiple-dose, parallel trial with a total duration of up to 50 days. The trial population will consist of healthy volunteers. Eligible subjects will be randomized to receive either subcutaneous (SC) apraglutide or matching placebo. The effect of apraglutide on gastric emptying of liquids will be assessed by the measure of PK of acetaminophen mixed with a liquid meal.

There will be two treatment periods, occurring according to the same sequence. In Period 1 acetaminophen will be given on Day 1, apraglutide/placebo will be injected on Day2. In Period 2 apraglutide/placebo will be injected on Day 9 and acetaminophen will be given on Day 10. This will allow to assess the PK of acetaminophen without the effect of apraglutide in Period 1, and to assess the PK of acetaminophen at the maximum concentration of apraglutide in Period 2.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 45 years inclusive
* Subjects who are willing and able to comply with the study procedures
* Subjects able to understand and willing to sign the informed consent
* Body mass index (BMI) of ≥18.0 to ≤30.0 kg/m2; and a total body weight of >50 kg (110 lb).
* Women of childbearing potential (WOCBP) having undergone bilateral tubal occlusion or with vasectomized partner. Sterilized or infertile or postmenopausal females.
* Male subjects with a WOCBP partner using highly effective methods of contraception and agreeing on no sperm donation during the trial and for 2 weeks after (EOT) visit.

Exclusion Criteria:

* History of clinically significant GI, bronchopulmonary, neurological, cardiovascular, endocrine, or allergic disease
* Known hypersensitivity to the investigational medicinal product (IMP), any of their excipients or drugs of the same class
* If capable of reproduction, unwilling to use an effective form of contraception
* If a WOCBP, a positive urine/blood pregnancy test
* Breast-feeding women
* Positive urine/blood test for alcohol and drugs of abuse
* Use of prohibited medications or herbal remedies
* Known presence or history of intestinal polyps
* Known presence or history of any type of cancer
* Pancreatic events such as acute pancreatitis, pancreatic duct stenosis, pancreas infection, and increased blood amylase and lipase (>2.0-5.0×upper limit of normal range)
* Participation in an investigational drug or device study within 30 days prior to Screening
* Donation of blood over 500 mL within 2 months prior to Screening
* Use of tobacco products (i.e., smokes more than 5 cigarettes per day or equivalent)
* Concomitant disease or condition that could interfere with, or for which the treatment of might interfere with, the conduct of the study, or that would, in the opinion of the Investigator, pose an unacceptable risk to the subject in this trial
* Any intercurrent clinically significant illness in the previous 28 days before Day 1 of this study
* Positive blood screen for human immunodeficiency virus (HIV) antigen/antibody combo, hepatitis A (HAV IGM), hepatitis B surface antigen (HBsAgB), or hepatitis C virus (HCV)
* Unwillingness or inability to comply with the study protocol for any other reason

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2023-03-02 (Actual); Primary Completion 2023-07-24 (Actual); Study Completion 2023-07-24 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) of acetaminophen | 0-300 Minutes
Time at which the maximum plasma concentration is observed (tmax) of acetaminophen | 0-300 Minutes
Area under the acetaminophen concentration-time curve: AUCinf (AUClast in case AUCinf cannot be estimated) | 0-14 hours
Area under the acetaminophen concentration-time curve: AUC0-300min | 0-300 Minutes
Area under the acetaminophen concentration-time curve: AUC0-60min | 0-60 Minutes

SECONDARY OUTCOMES:
Height | Through study completion, up to 24 days
  In cm
Weight | Through study completion, up to 24 days
  In kg
Physical examination | Through study completion, up to 24 days
  Clinically significant outcome (as normal or abnormal) for physical examination of eyes, neurological, gastrointestinal, respiratory, circulatory, muscular, cardiovascular, lymphatic, ears, nose, throat.
The incidence, nature and severity of adverse events (AEs) with apraglutide | Through study completion, up to 24 days
Clinical chemistry | Through study completion, up to 24 days
  Clinical Chemistry panel of analytes will be examined for clinically significant changes.
  Clinical chemistry analytes will be listed by subject. Descriptive statistics will be used to assess any changes in clinical laboratory results during and following trial treatment administration. Values outside the reference ranges will be highlighted and clinical significance stated.
Hematology | Through study completion, up to 24 days
  Hematology panel of analytes will be examined for clinically significant changes.
  Hematology analytes will be listed by subject. Descriptive statistics will be used to assess any changes in clinical laboratory results during and following trial treatment administration. Values outside the reference ranges will be highlighted and clinical significance stated.
Hemostasis | Through study completion, up to 24 days
  Hemostasis INR will be examined for clinically significant changes
Anti-drug antibodies (ADA) analysis | Through study completion, up to 24 days
  ADA will be will be examined for clinically significant changes
Urine analysis | Through study completion, up to 24 days
  Urine analysis panel of analytes will be examined for clinically significant changes
Occurrence of clinically relevant changes in vital signs | Through study completion, up to 24 days
  Systolic and diastolic blood pressure in mmHg
Occurrence of clinically relevant changes in vital signs | Through study completion, up to 24 days
  Pulse rate in Beats per Minute
Changes in body temperature in °C | Through study completion, up to 24 days
Occurrence of clinically relevant changes in electrocardiogram | Through study completion, up to 24 days
  ECG QT Interval
Occurrence of clinically relevant changes in electrocardiogram | Through study completion, up to 24 days
  ECG PR interval
Occurrence of clinically relevant changes in electrocardiogram | Through study completion, up to 24 days
  ECG QRS interval
Occurrence of clinically relevant changes in electrocardiogram | Through study completion, up to 24 days
  ECG rhythm

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz Masior, Study Director — VectivBio AG
Locations (1):
- ICON Clinical Research Unit, Groningen, Netherlands